CLINICAL TRIAL: NCT06027502
Title: Cardioprotective Benefit of Passive Heat Therapy in Higher-Level Spinal Cord Injury: Safety and Proof of Concept
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, James Laskin, Adjunct Profesor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H22-03599
Record Dates: First submitted 2023-07-30; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Spinal Cord Injuries; Cardiovascular Diseases; Health Behaviour; Physical Inactivity
Keywords: Spinal cord injury; Passive heating; Exercise response; Cardio protection
MeSH Terms: conditions — Spinal Cord Injuries; Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Two groups, those with a cervical level SCI and a control group of non-disabled healthy individuals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Passive Heating (Experimental): Passive heating will be achieved by approximately 45 min of immersion in a Hot Tub at 40 degrees celsius
  Interventions: Behavioral: Passive Heating

INTERVENTIONS:
Behavioral: Passive Heating — 20 minutes of baseline data collection, up to 45 minutes of immersion in the hot tub to achieve a core temperature of 38.5 degrees celsius, followed by up to 90 minutes of recovery.

SUMMARY:
As compared to the general population, those living with a spinal cord injury (SCI) are at a greater risk of cardiovascular (CV) diseases.The investigators know that regular exercise can help lessen the risk of CV diseases. However, those with higher level SCI have a limited ability to exercise due to their loss of function. Heat therapy has been shown to promote significant health benefits in populations with health challenges and has demonstrated a mild exercise like response. The investigators aim to extend these findings and develop a practical passive heat therapy program appropriate for safe home use.

DETAILED DESCRIPTION:
The risk of cardiovascular diseases for people with a spinal cord injury (SCI) is approximately 3x greater than the general population, and Cardiovascular (CV) diseases account for ~40% of deaths in SCI. Traditional CV risk factors are unable to fully explain these outcomes. This group also has other secondary complications that are concerning, including susceptibility to infections and metabolic health issues. Some of the increased risk in SCI is due to a relatively sedentary lifestyle and insufficient exercise capability. This is particularly insidious in those living with tetraplegia with poor cardiovascular responses to exercise or even the inability to exercise due to upper limb paralysis.

Heat therapy in the form of hot baths and saunas has been utilized for centuries, with common reports of improved quality of life and overall improved well-being. A 20-year prospective study on 2,315 middle-aged men (at enrolment) in Finland reported that regular sauna bathing was associated with reduced risk of sudden cardiac death, coronary heart disease, CV disease, and all-cause mortality. Further, more frequent sauna bathing sessions were related to a considerably decreased risk of fatal cardiac and CV events, as well as all-cause mortality independently from conventional risk factors, activity levels, and diet. The mechanisms which underlie these improvements remain largely unknown. It has been proposed that CV benefits of exercise training are partly mediated by repeated increases in core temperature. Exercise and heat stress elicit many common physiological responses, including increases in core temperature, heart rate and contractility, redistribution of blood flow, and changes in conduit vessel endothelial shear stress, all of which are believed to improve CV health. Additionally, heat exposure and exercise induce the expression of heat shock proteins, which stabilize a variety of other proteins that reduce vascular inflammation and oxidative stress, improve NO bioavailability, promote angiogenesis, and improve glucose signaling.

SCI results in a host of physiological changes that greatly increase CV risk and vascular dysfunction following injury. Increased arterial stiffness and vascular resistance are common features in SCI, likely secondary to the loss of sympathetic innervation below the lesion, increased circulating vasoconstrictors, and subsequent oxidative stress and vascular inflammation. Heat exposure is a stress to the CV system, like exercise, which may result in numerous chronic adaptations that improve vascular and metabolic function, resulting in a profoundly reduced risk of CV disease.

Passive heat therapy may provide a novel and practical approach to help these individuals. There have been observed profound improvements in vascular and metabolic function as well as indications of benefits to the immune system and reductions in inflammation in healthy but sedentary able-bodied people after long-term passive heat exposure. Similar benefits were observed in obese women with polycystic ovary syndrome. Recent studies in SCI with lower limb and full-body (only in low level SCI) immersion have demonstrated the potential of hot water immersion to be safe, with the potential to stimulate a cardio-protective response. The proposed pilot study is the first step in developing a unique approach for combating CV dysfunction in the SCI population.

Specifically, the goal of this pilot study is to build on the current literature and demonstrate the safety, tolerance, and effectiveness (providing a mild/moderate exercise response) of a ~ 45-minute full-body hot water immersion in those with higher level SCI (T7-C4). Ultimately, the investigators will develop a protocol for translating these and future findings to the home environment and use of a typical bathtub, thereby demonstrating that passive heat therapy is a viable approach to improve health in the SCI population.

Water immersion is the preferred method of heating since it is capable of increasing core temperature and heart rate at a rate similar to moderate-intensity exercise. It is difficult to achieve increases in core temperature solely via air convection, including in paraplegic SCI, as participants rapidly acclimate to the heat with increased sweating, limiting the rise in core temperature and heart rate. In addition, hot tubs, whirlpools, and baths are available in the community, and most should provide wheelchair access. In addition, a water bath in the home is an acceptable alternative to a hot tub to sufficiently raise core body temperature. Furthermore, water is an excellent conductor of heat, and will provide uniform heating across the participants' body. This helps eliminate "hot spots" that could result in a burn, particularly in insensate areas of skin.

For this study, up to 16 individuals will be recruited from International Collaboration on Repair Discoveries (ICORD) Physical Activity Research Centre (PARC) Community as well as from the larger SCI community who live with a T7-C4 injury. In addition, the investigators will be recruiting up to 6 control participants who are otherwise healthy individuals who do not live with an SCI. During the single, approximately 45-minute exposure to this passive heating modality the investigators will be measuring heart rate, blood pressure (mean arterial pressure), cardiac output, respiration rate and core temperature. This descriptive study will have each participant attend the lab for a single session.

After a 20 min of baseline data collection period the participant will be transferred to the hot tub using a standard Hoyer lift and sling. While in the hot tub they will remain in a semi-reclined position. Initially the participant will be submersed up to the clavicular level with one arm out of water until the core temperature reaches 38.5 C (about 20 - 25 minutes), once this temperature has been reached, they will be positioned so that the water level lays between the waist and mid-sternum. The water level on the participant's body will be adjusted such that a core temperature of 38.5 C for 20 minutes (typical moderate exercise duration) is maintained. If the participants core temperature exceeds 39.5 C the session will be terminated and the participant removed from the hot tub. While in the hot tub the participant may drink water ad lib with the volume recorded.

While submersed in the hot tub:

* Core temperature, blood pressure, blood flow, and heart rate will be monitored continuously
* Oxygen consumption will be assessed every 5 minutes
* Cardiac output will be assessed every 10 minutes

Once the ~45 min of immersion has been completed the participant will be removed from the hot tub using the Hoyer lift and placed back on the plinth in a semi-reclined position for 20 minutes of recovery/rest. While in this recovery position core temperature, blood pressure, blood flow, and heart rate will be monitored continuously.

After this initial recovery period the investigators will assist the participant as necessary to help the participant get dressed, weighed, testing equipment removed and will continue resting comfortably in the participant's everyday wheelchair for 60-90 min.

The outcome variables to be examined include the following:

* Heart rate
* Blood pressure (systolic, diastolic, mean arterial pressure, beat to beat)
* Core temperature (via CorTemp© "smart pill and Bear Hugger)
* Cardiac output
* Oxygen consumption
* Brachial and cerebral artery blood flow
* End tidal gas - respiration rate
* Weight loss

Each of the outcome variables will be examined in both an individual and pooled manner (average and standard deviation). In addition, any potential group trends (e.g., injury level [thoracic versus cervical] and severity [ American Spinal Injury Association Impairment Scale (AIS) score]) in terms of the response to the passive heating stimulus will be examined.

ELIGIBILITY:
Inclusion Criteria:

* sedentary to active individuals living with a spinal cord injury and have injury level between T7 and C4 (of any AIS level)*
* at least 2 years post-injury*
* be able to do a level transfer with minimal assistance*
* engaged in a regular and consistent bowel/bladder management program*
* be 19 years of age or older
* be able to communicate effectively in English
* If present, self-reported well controlled/predictable orthostatic hypertension and/or autonomic dysreflexia*
* be fully vaccinated against COVID-19 (initial 2 doses and 1 booster)

  * these criteria do not apply to the non-SCI controls

Exclusion Criteria:

* smoke/use tobacco products
* have any cardiac/respiratory illness or diabetes mellitus
* known diverticulitis
* hypertensive (Systolic Blood Pressure >140 mmHg and/or Diastolic Blood Pressure >190 mmHg)
* scheduled MRI investigation in the 7 days following the data collection session
* take prescription medications that affect blood vessels, other than contraceptives
* have used an erectile dysfunction related medication (e.g., Viagra or Cialis) in the past 48 hours
* have unhealed fracture, or contracture, that would interfere with a simple chair to tub transfer and/or donning/doffing clothing
* have an unhealed pressure sore of any grade and/or open skin areas
* have unstable medical/psychiatric condition or substance abuse disorder that is likely to affect their ability to complete this study
* have underlying health conditions or injuries that would impact their ability to tolerate a mild exercise response or hot water immersion
* have uncontrolled orthostatic hypotension i.e., blood pressure does not return to normal within 2-3 minutes after standing or transferring*
* have underlying health conditions that put them at greater risk for COVID-19 (e.g., respiratory illness, compromised immunity, or chronic health condition)
* have any COVID-19 related symptoms (e.g., new or worsening cough, shortness of breath, sore throat, runny nose or nasal congestion, hoarse voice, difficulty swallowing, new smell or taste disorders, nausea, vomiting, diarrhea, abdominal pain, unexplained fatigue, chills or headache)
* have a fever
* have travelled outside Canada or had close contact with anyone who has travelled outside Canada in the past 14 days
* have close contact with anyone with respiratory illness or a confirmed or probable case of COVID-19
* are currently self-isolating

  * these criteria do not apply to the non-SCI controls

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Core temperature | Continuously recorded - Baseline (Pre immersion - 20 minutes), Immersion (45 minutes) and Post-immersion/Recovery (60 to 90 minutes)
  As measured by CorTemp smart pill and the Bair Hugger system
Oxygen consumption | Recorded every 5 minutes -Baseline (Pre immersion - 20 minutes), Immersion (45 minutes) and Post-immersion/Recovery (60 to 90 minutes)
  As measured by open circuit spirometer
Cardiac output | Recorded every 5 minutes -Baseline (Pre immersion - 20 minutes), Immersion (45 minutes) and Post-immersion/Recovery (60 to 90 minutes)
  As measured indirectly by Finopres©
Blood pressure | Continuously recorded - Baseline (Pre immersion - 20 minutes), Immersion (45 minutes) and Post-immersion/Recovery (60 to 90 minutes)
  As measured indirectly by Finopres©
Heart rate | Continuously recorded - Baseline (Pre immersion - 20 minutes), Immersion (45 minutes) and Post-immersion/Recovery (60 to 90 minutes)
  As measured indirectly by Finopres©

SECONDARY OUTCOMES:
Cerebral artery blood flow | Recorded every 5 minutes -Baseline (Pre immersion - 20 minutes), Immersion (45 minutes) and Post-immersion/Recovery (60 to 90 minutes)
  As measured by arterial doppler ultrasound
Brachial arterial blood flow | Recorded every 5 minutes -Baseline (Pre immersion - 20 minutes), Immersion (45 minutes) and Post-immersion/Recovery (60 to 90 minutes)
  As measured by arterial doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: James J Laskin, PT,PhD, Principal Investigator — Department of Occupational Science & Occupational Therapy, UBC
Locations (1):
- ICORD Blusson SPinal Cord Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunt VE, Howard MJ, Francisco MA, Ely BR, Minson CT. Passive heat therapy improves endothelial function, arterial stiffness and blood pressure in sedentary humans. J Physiol. 2016 Sep 15;594(18):5329-42. doi: 10.1113/JP272453. Epub 2016 Jun 30. PMID 27270841
- [Result] Larson EA, Ely BR, Francisco, MA, Brunt VE, Minson CT. Thermoregulatory Response to Acute Passive Heat Exposure in Individuals with Low-level Spinal Cord Injury. FASEB J. 2019;33(1):838.19.
- [Result] Gass EM, Gass GC. Thermoregulatory responses to repeated warm water immersion in subjects who are paraplegic. Spinal Cord. 2001 Mar;39(3):149-55. doi: 10.1038/sj.sc.3101117. PMID 11326325
- [Result] Brunt VE, Eymann TM, Francisco MA, Howard MJ, Minson CT. Passive heat therapy improves cutaneous microvascular function in sedentary humans via improved nitric oxide-dependent dilation. J Appl Physiol (1985). 2016 Sep 1;121(3):716-23. doi: 10.1152/japplphysiol.00424.2016. Epub 2016 Jul 14. PMID 27418688